CLINICAL TRIAL: NCT07248696
Title: Tislelizumab Plus Chemotherapy With Response-Adapted Radiotherapy for de Novo Metastatic Nasopharyngeal Carcinoma: A Prospective, Phase II Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xin Zhang, Associate Chief Physician, Chongqing University Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Daybreak-01
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: nasopharyngeal carcinoma; de novo metastatic; tislelizumab
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- response-adapted radiotherapy (Experimental): This is a prospective phase II study that enrolled patients with previously untreated de novo metastatic nasopharyngeal carcinoma who achieved either a complete response (CR) or partial response (PR) after 4-6 cycles of treatment with gemcitabine plus cisplatin (GP regimen) chemotherapy combined with tislelizumab. Based on tumor response stratification, these patients received locoregional radiotherapy and radiotherapy for metastatic lesions, followed by sequential tislelizumab maintenance therapy.
  Interventions: Radiation: response-adapted radiotherapy

INTERVENTIONS:
Radiation: response-adapted radiotherapy — Induction Treatment Regimen:
  • Tislelizumab+Gemcitabine+Cisplatin for 4-6 cycles .
  Response-Adapted Radiotherapy:
  * Patients achieving CR after induction therapy require no radiotherapy.
  * Patients achieving PR after induction therapy: Radiotherapy (55 Gy/20 fractions, 5 fractions per week, over 4 weeks) to the residual primary nasopharyngeal lesion and metastatic cervical lymph nodes. Radiotherapy for metastatic lesions concurrently or sequentially with locoregional radiotherapy.
  Immunotherapy Regimen:
  maintenance therapy with tislelizumab monotherapycontinues until disease progression, unacceptable toxicity, or withdrawal of consent, whichever occurs first. The total treatment duration shall not exceed 2 years

SUMMARY:
This study is aimed to evaluate the efficacy and safety of tislelizumab combined with chemotherapy and response-adapted radiotherapy in patients with de novo metastatic nasopharyngeal carcinoma

DETAILED DESCRIPTION:
This is a prospective phase II study that enrolled patients with previously untreated de novo metastatic nasopharyngeal carcinoma who achieved either a complete response (CR) or partial response (PR) after 4-6 cycles of treatment with gemcitabine plus cisplatin (GP regimen) chemotherapy combined with tislelizumab. Based on tumor response stratification, these patients received locoregional radiotherapy and radiotherapy for metastatic lesions, followed by sequential tislelizumab maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years.
2. Newly diagnosed nasopharyngeal carcinoma with pathological confirmation of non-keratinizing carcinoma (WHO type II or III).
3. Stage IV (T1-4N0-3M1a and M1b) according to the AJCC/UICC 9th edition clinical staging system for NPC.
4. Achieved complete response (CR) or partial response (PR) by imaging evaluation after 4-6 cycles of GP chemotherapy combined with tislelizumab.
5. ECOG performance status: 0-1.
6. Adequate organ function.

Exclusion Criteria:

1. Recurrent or metastatic nasopharyngeal carcinoma after radical treatment.
2. Other malignancies diagnosed or treated within the past 5 years (except basal cell carcinoma, cervical carcinoma in situ, and superficial bladder tumors).
3. Previous treatment with immune checkpoint inhibitors.
4. Pregnancy or lactation (consider pregnancy testing for women of childbearing age and emphasize effective contraception during treatment).
5. Active or history of autoimmune diseases.
6. Concurrent medical condition requiring the use of immunosuppressive medications.
7. Active hepatitis B or C infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-04 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 1-year
  PFS is defined as the time from the initiation of treatment until the first occurrence of locoregional progression, distant metastatic progression, or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
OS | 1-year
Local Regional Control | 1-year
Distant Metastasis Control | 1-year
ORR | 1-year
DoR | 1-year

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Due to ethical requirements, the data can be obtained via email.

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, et al. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021;71(3):209-249. 2. Ng SH, Chan SC, Yen TC, et al. Pretreatment evaluation of distant-site status in patients with nasopharyngeal carcinoma: accuracy of whole-body MRI at 3-Tesla and FDG-PET-CT. Eur Radiol. 2009;19(12):2965-2976. 3. Zou X, You R, Liu H, et al. Establishment and validation of M1 stage subdivisions for de novo metastatic nasopharyngeal carcinoma to better predict prognosis and guide treatment. Eur J Cancer. 2017;77:117-126. 4. Zhang L, Huang Y, Hong S, et al. Gemcitabine plus cisplatin versus fluorouracil plus cisplatin in recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 trial. Lancet. 2016;388(10054):1883-1892. 5. Yang Y, Pan J, Wang H, et al. Tislelizumab plus chemotherapy as first-line treatment for recurrent or metastatic nasopharyngeal cancer: A multicenter phase 3 trial (RATIONALE-309). Cancer Cell. 2023;41(6):1061-1072 e1064. 6. Mai HQ, Chen QY, Chen D, et al. Toripalimab Plus Chemotherapy for Recurrent or Metastatic Nasopharyngeal Carcinoma: The JUPITER-02 Randomized Clinical Trial. JAMA. 2023;330(20):1961-1970. 7. Yang Y, Qu S, Li J, et al. Camrelizumab versus placebo in combination with gemcitabine and cisplatin as first-line treatment for recurrent or metastatic nasopharyngeal carcinoma (CAPTAIN-1st): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2021;22(8):1162-1174. 8. You R, Liu YP, Huang PY, et al. Efficacy and Safety of Locoregional Radiotherapy With Chemotherapy vs Chemotherapy Alone in De Novo Metastatic Nasopharyngeal Carcinoma: A Multicenter Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020;6(9):1345-1352. 9. Chen SY, Duan XT, Li HF, et al. Efficacy of sequential chemoradiotherapy combined with toripalimab in de novo metastatic nasopharyngeal carcinoma: A phase II trial. Cell Rep Med.